CLINICAL TRIAL: NCT05689333
Title: A Prospective, Single-arm, Non-comparative, Open-label, Monocular, Post Approval Study to Assess Safety and Device Performance of the Vista Vitrectomy Probe During Vitrectomy Surgery
Brief Title: A Study to Evaluate the Safety and Performance of the Vista Probe for Vitrectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VISTA Ophthalmics (Industry)
Collaborators: CBCC Global Research (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBCC/2022/009
Record Dates: First submitted 2022-12-22; First posted 2023-01-19 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Vitrectomy
Keywords: Vitrectomy Probe; Vitreous aspiration & cutting; Dissect tissue in the eye

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- 27 GA Vista Ophthalmics vitrector (Experimental): The vitrectomy will be performed through the pars plana using the 27 GA Vista Ophthalmics vitrector.
  Interventions: Device: Vista Vitrectomy Probe

INTERVENTIONS:
Device: Vista Vitrectomy Probe — Vitrectomy will be performed through 27 GA Vista Ophthalmics vitrector

SUMMARY:
This is a prospective, single-arm, non-comparative, open-label, monocular, post approval study to assess safety and device performance of the Vista Vitrectomy Probe during vitrectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant with age ≥ 18 years at the time of screening.
* Subject must have a clinical indication for anterior vitrectomy.
* Subjects must be able to understand and voluntarily provide written informed consent before screening, following an explanation of the nature and purpose of this study.
* Subjects must be willing and able to comply with all treatment and follow-up study procedures.

Exclusion Criteria:

* Subjects who have experienced any significant trauma in the operative eye within the past month.
* Subjects with any active ocular infection or history of any herpetic infection that has cleared less than one month prior to the pre-operative visit.
* Subjects with prior history of uncontrolled glaucoma or uveitis refractory to treatment or ocular hypertension (IOP>30mm Hg) in study eye.
* Subjects with any medical condition (e.g., uncontrolled diabetes) that, based on the Investigator's medical judgment, poses a concern for the subjects' safety.
* Female subjects of child bearing potential with positive urine pregnancy test
* Subjects who have participated in any drug or device clinical investigation within 30 days prior to entry into or during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Incidence of post-operative rates of retinal tears | Month 1
  Calculate the incidence of post-operative rates of retinal tears
Incidence of retinal detachment | Month 1
  Calculate the incidence of post-operative retinal detachment
Incidence of sclerotomy complications like leakage | Month 1
  Calculate the incidence of post-operative sclerotomy complications like leakage
Incidence of ocular hypotony | Month 1
  Calculate the incidence of post-operative ocular hypotony
Incidence of choroidal detachment | Month 1
  Calculate the incidence of post-operative choroidal detachment
Incidence of visually significant vitreous hemorrhage | Month 1
  Calculate the incidence of post-operative visually significant vitreous hemorrhage (visual acuity defined by counting fingers or worse)
Incidence of endophthalmitis | Month 1
  Calculate the incidence of post-operative endophthalmitis

SECONDARY OUTCOMES:
Surgeon- will assess device adequacy for removal of vitreous | Day 0 (Operative Visit)
  Surgeon-assess device adequacy for removal of vitreous will be summarized using counts and percentages
Percentage of eyes with clinical evidence of incomplete vitrectomy, such as vitreous strands or pupil peaking | Days1, 7, 30 & 90
  Percentage of eyes with clinical evidence of incomplete vitrectomy, such as vitreous strands or pupil peaking, at any post-operative visit will be summarized using counts and percentages

CONTACTS AND LOCATIONS:
Overall Officials: Don Knowles, Study Chair — VISTA Ophthalmics
Locations (4):
- United States (4):
  - CBCC Global Research Site:003, Los Angeles, California
  - CBCC Global Research Site:002, Bradenton, Florida
  - CBCC Global Research Site:001, Bala-Cynwyd, Pennsylvania
  - CBCC Global Research Site:004, McAllen, Texas